CLINICAL TRIAL: NCT00823862
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled Dose-Escalation Study of SD-101 to Assess the Safety, Pharmacodynamics, and Preliminary Evidence of Anti-Viral Effect in Subjects Diagnosed With Chronic Hepatitis C, Genotype 1
Brief Title: Safety Study of SD-101 (a Novel C Type Toll-like Receptor 9 (TLR9) Agonist) for the Treatment of Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: Synteract, Inc. (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DV3-HCV-01; 2008-001708-22 (EudraCT Number)
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Immunostimulatory sequence (ISS); TLR9 (toll-like receptor 9); interferon (IFN); ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (SD-101) (Experimental): SD-101 in cohorts of escalating doses
  Interventions: Drug: SD-101; Drug: ribavirin

INTERVENTIONS:
Drug: SD-101 — Intramuscular (IM)
  Other Names: CpG Class C Immunostimulatory Sequence (ISS); TLR9 Agonist
Drug: ribavirin — oral, 2 times per day, for 2 months

SUMMARY:
To determine safety, tolerability, and preliminary efficacy of escalating doses of SD-101 alone and SD-101 plus ribavirin in subjects with chronic hepatitis C and no prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written, informed consent
* Male or female subjects, 18 to 55 years of age.
* Subject must have chronic infection HCV, genotype 1.
* Serum HCV-RNA concentrations 100,000 IU/mL to 10,000,000 IU/mL
* No prior treatment for HCV.
* Must be negative for hepatitis B (HBV) and human immunodeficiency virus (HIV).
* Must be willing to use dual method of contraception (i.e., barrier and spermicide; birth control pills and barrier) during the study.
* No known hypersensitivity to study medication or to drugs chemically related to the study.

Exclusion Criteria:

* Prior treatment with IFN-based therapies and/or anti-viral therapies.
* Women with ongoing pregnancy or breast feeding and male partners of women who are pregnant.
* Reduced kidney function.
* Presence of concomitant liver diseases
* Signs or symptoms of hepatocellular carcinoma.
* Thyroid disease currently poorly controlled on prescribed medications.
* History of hemoglobinopathy.
* Evidence of severe retinopathy.
* Other serious medical conditions, including human immunodeficiency virus, cancer (excluding non-melanoma skin cancer), or evidence of drug or alcohol abuse.
* Subjects with documented or presumed coronary artery disease, pulmonary disease, or cerebrovascular disease
* Clinically significant acute or chronic illnesses.
* History of severe psychiatric disease, especially depression, characterized by a suicide attempt, hospitalization for psychiatric disease, or a period of disability as a result of psychiatric disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Adverse event timing, duration, and severity. | Between doses and up to 3 months after last dose

SECONDARY OUTCOMES:
Biomarker analysis of blood sample | pre and 24 hour post dose
Viral load in blood sample | each visit

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Cianciara, MD, Principal Investigator — Warszawski Uniwersytet Medyczny
Locations (5):
- Poland (5):
  - Klinika Chorób Zakaźnych i Hepatologii Collegium Medicum Uniwersytet Mikołaja Kopernika, Bydgoszcz
  - Katedra i Klinika Chorób Zakaźnych Uniwersytet Medyczny w Lublinie, Lublin
  - Wojewódzki Szpital Zakaźny - Klinika Hepatologii i Nabytych Niedoborów Immunologicznych, Warsaw
  - Wojewódzki Szpital Zakaźny, Warsaw
  - EMC Instytut Medyczny S.A. Szpital Specjalistyczny z Przychodnią "EuroMediCare", Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided
3/2017 no change to status in this Phase 1 study